CLINICAL TRIAL: NCT00663936
Title: A Phase 2a Multi-center, Randomized, Double Blind, Placebo-controlled Study to Investigate the Efficacy and Safety of T-817MAa in Patients With Mild to Moderate Alzheimer's Disease
Brief Title: Efficacy and Safety of T-817MA in Patients With Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: FUJIFILM Toyama Chemical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AA4437420
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2012-12

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; Alzheimer's
MeSH Terms: conditions — Alzheimer Disease | interventions — 1-(3-(2-(1-benzothiophen-5-yl) ethoxy) propyl)-3-azetidinol maleate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): T-817MA once daily
  Interventions: Drug: T-817MA
- 2 (Placebo Comparator): Placebo once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: T-817MA — 224 mg T-817 MA once daily
  Arms: 1
Drug: Placebo — Placebo once daily
  Arms: 2

SUMMARY:
The primary objective of the study is to evaluate the efficacy of T-817MA in AD patients to treat dementia. Efficacy will be cognitive function, as measured by the ADAS-cog cognitive assessment.

The secondary objectives of the study are to evaluate the safety of T-817MA and the activities of daily living (assessed with the ADCS-ADL) of AD patients taking T-817MA, and to evaluate the efficacy of T-817MA in AD patients with an overall global assessment using the ADCS-CGIC.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female (post-menopausal or surgically sterile)
2. Patients with Mild to moderate Alzheimer's disease who are receiving Donepezil.
3. Age 50 to 90 inclusive
4. Patients must be living in the community
5. Patients must have an eligible informant or study partner (caregiver)
6. Patients and eligible informant or study partner (caregiver) must be able to read and understand English.
7. Informed consent obtained from both the patient and the caregiver etc (According to the protocol)

Exclusion Criteria:

1. Patients with clinically significant cardiac, hepatic or renal impairment
2. Patient have a dementia not of the Alzheimer's type etc (According to the protocol)
3. Patients who are taking any drug other than donepezil for Alzheimer's disease, including rivastigmine (Exelon®), galantamine (Razadyne®), memantine (Namenda™) or tacrine (Cognex®) taken within twelve (12) weeks of the Baseline Visit (Visit 2).

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 373 (Actual)
Dates: Start 2008-04; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of the efficacy of T-817MA in AD patients to treat dementia. Efficacy will be cognitive function, as measured by the ADAS-cog cognitive assessment. | 52 weeks

SECONDARY OUTCOMES:
Secondary objectives are to evaluate the safety of T-817MA and the activities of daily living (ADCS-ADL) of AD patients taking T-817MA, and to evaluate the efficacy of T-817MA in AD patients with an overall global assessment using the ADCS-CGIC. | 52 weeks

CONTACTS AND LOCATIONS:
Locations (35):
- United States (33):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Northwest NeuroSpecialists, Tucson, Arizona
  - Collaborative Neuroscience Network, Inc., Garden Grove, California
  - Southwest Institute for Clinical Research, Inc., Rancho Mirage, California
  - Pacific Research Network, Inc., San Diego, California
  - San Francisco Clinical Research Center, San Francisco, California
  - Radiant Research, Denver, Colorado
  - Geriatric and Adult Psychiatry, LCC, Hamden, Connecticut
  - Research Center for Clinical Studies, Inc., Norwalk, Connecticut
  - NeuroPsychiatric Center of the Palm Beaches, Boynton Beach, Florida
  - Galiz Research, Miami Springs, Florida
  - Anchor Research Center, Naples, Florida
  - Renstar Medical Research, Ocala, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - Johnnie B. Byrd Sr. Alzheimer's Center and Research Institute, Tampa, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Columbus Research & Wellness Institute, Columbus, Georgia
  - Agewell, Indianapolis, Indiana
  - Cleveland Clinic - Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - Comprehensive Clinical Research, Berlin, New Jersey
  - Memory Enhancement Center of America, Toms River, New Jersey
  - Brooklyn Medical Institute, Brooklyn, New York
  - SPRI Clinical Trials, Brooklyn, New York
  - Alzheimer's Disease Center, U. of Rochester Medical Center, Rochester, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - The Alzheimer's Memory Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Clinical Trials of America, Inc., Winston-Salem, North Carolina
  - The Clinical Trials Center, Jenkintown, Pennsylvania
  - CRI Worldwide, LLC, Philadelphia, Pennsylvania
  - Innovative Clinical Trials, San Antonio, Texas
  - IPC Research, Waukesha, Wisconsin
- Canada (2):
  - St. Joseph's Hospital, Saint John, New Brunswick
  - Toronto Memory Program, Toronto, Ontario